CLINICAL TRIAL: NCT03903874
Title: Testing Scalable, IVR-supported Cancer Prevention Interventions in the Rural Alabama Black Belt
Acronym: DIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Dorothy Pekmezi, PhD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-300003238; R01CA233550 (NIH)
Record Dates: First submitted 2019-03-31; First posted 2019-04-04 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: assessment staff will be blind to condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DIAL intervention (Experimental): Deep south Interactive voice response system Active Lifestyle (DIAL) intervention. Participants will receive 12 months of automated physical activity phone counseling. Participants will report their physical activity to the IVR system each day for 3 months, twice/week in months 3-6, and once/week in months 6-12 and receive progress feedback via IVR system, along with community health worker support.
  Interventions: Behavioral: Deep south Interactive voice response system supported Active Lifestyle (DIAL)
- Wait List Control (No Intervention): The wait list control participants will be instructed to maintain their normal routine until completion of the 6-month assessments and then receive the same 12-month DIAL intervention. To maintain engagement, these participants will be involved in monthly lunch and learns, focus groups, etc on cancer topics other than PA (e.g., screening) during the wait period.

INTERVENTIONS:
Behavioral: Deep south Interactive voice response system supported Active Lifestyle (DIAL) — 12 months of automated telephone physical activity counseling with community health worker support
  Arms: DIAL intervention

SUMMARY:
This protocol involves a randomized controlled trial (N=240) to test the efficacy of the Deep south Active Lifestyle (DIAL intervention) telephone-based physical activity counseling intervention vs. a wait list condition. Assessments of MVPA and psychosocial variables will occur at baseline, 6, 12, and 18 months. Primary aim. Test the efficacy of DIAL intervention vs. wait list control. Hypotheses are that the participants receiving DIAL intervention will report significantly greater increases in MVPA (based on 7-Day Physical Activity Recalls, accelerometers) from baseline to 6 and 12 months than the wait list control arm. Exploratory Aims. Examine 1) Intervention effects on physical performance and psychosocial variables (anxiety, depression, fatigue, sleep disturbance; corroborate self report sleep improvements from pilot with accelerometry); 2) Changes in MVPA from 12-18 months to assess long term (6 months post-intervention) maintenance in the intervention arm and ascertain replicability of intervention effects in wait list control arm; 3) Intervention costs; 4) Potential mediators (social support from family, friends, CHAs, theoretical constructs directly targeted by the intervention) and moderators (education, neighborhood/environmental features) of treatment efficacy; 5) Potential barriers/ facilitators to widespread implementation of DIAL intervention in rural Black belt counties by Deep South Network for Cancer Control.

DETAILED DESCRIPTION:
This protocol involves a randomized controlled trial (N=240) to test the efficacy of the Deep south Active Lifestyle (DIAL intervention) telephone-based physical activity counseling intervention vs. a wait list condition. Assessments of MVPA and psychosocial variables will occur at baseline, 6, 12, and 18 months.

Primary aim. Test the efficacy of DIAL intervention vs. wait list control. Hypotheses are that the participants receiving DIAL intervention will report significantly greater increases in MVPA (based on 7-Day Physical Activity Recalls, accelerometers) from baseline to 6 and 12 months than the wait list control arm.

Exploratory Aims. Examine 1) Intervention effects on physical performance and psychosocial variables (anxiety, depression, fatigue, sleep disturbance; corroborate self report sleep improvements from pilot with accelerometry); 2) Changes in MVPA from 12-18 months to assess long term (6 months post-intervention) maintenance in the intervention arm and ascertain replicability of intervention effects in wait list control arm; 3) Intervention costs; 4) Potential mediators (social support from family, friends, CHAs, theoretical constructs directly targeted by the intervention) and moderators (education, neighborhood/environmental features) of treatment efficacy; 5) Potential barriers/ facilitators to widespread implementation of DIAL intervention in rural Black belt counties by Deep South Network for Cancer Control.

ELIGIBILITY:
Inclusion Criteria:

* Insufficiently active (engaging in MVPA < 60 minutes per week)
* Residents of participating rural Black Belt counties (Dallas, Marengo, Choctaw, Sumter, Hale, Greene)
* BMI 18.5-45
* Able to speak and read English
* Willing to be randomized to either study arm and adhere to study protocol
* Able to regularly access a telephone (own a cell phone or work/home landline) to complete IVR calls

Exclusion Criteria:

* Serious medical conditions that would make physical activity unsafe (history of heart disease, myocardial infarction, angina, stroke, orthopedic conditions which limit mobility),
* Planning to move from the area within the next 18 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Pekmezi, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama At Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brown NI, Powell MA, Baskin M, Oster R, Demark-Wahnefried W, Hardy C, Pisu M, Thirumalai M, Townsend S, Neal WN, Rogers LQ, Pekmezi D. Design and Rationale for the Deep South Interactive Voice Response System-Supported Active Lifestyle Study: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 May 25;10(5):e29245. doi: 10.2196/29245. PMID 34032575

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DIAL intervention | Wait List Control
Started | 123 | 122
Completed | 108 | 110
Not Completed | 15 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DIAL intervention | Wait List Control | Total
Number analyzed (Participants) | 123 | 122 | 245
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 69 | 73 | 142
  >=65 years | 54 | 49 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.41 (14.25) | 59.27 (12.64) | 59.34 (13.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 110 | 223
  Male | 10 | 12 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 123 | 122 | 245
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 119 | 120 | 239
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 123 | 122 | 245

OUTCOME MEASURES:

1. Primary Outcome: Changes in Moderate-vigorous Intensity Physical Activity
Description: Changes in min/week of moderate-vigorous intensity physical activity from baseline to 6 months, based on 7-Day Physical Activity Recall interviews
Time Frame: baseline, 6 months, 12 months, 18 months
Population: intent to treat analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: min/week of physical activity
Arm/Group | DIAL intervention | Wait List Control
Number analyzed (Participants) | 123 | 120
min/week of physical activity | 67.35 [45.43 to 89.28] | 4.09 [-17.34 to 25.53]

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | DIAL intervention | Wait List Control
All-Cause Mortality (participants affected / at risk) | 1/123 | 0/122
Serious Adverse Events (participants affected / at risk) | 6/123 | 1/122
Other Adverse Events (participants affected / at risk) | 10/123 | 14/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DIAL intervention (N=123) | Wait List Control (N=122)
hospitalized (General disorders) | 1 (1) | 0 (0)
kidney transplant (Renal and urinary disorders) | 1 (1) | 0 (0)
bursitis, bulging disc; hand (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
high blood pressure, triple bypass, stroke (Cardiac disorders) | 2 (2) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DIAL intervention (N=123) | Wait List Control (N=122)
Back, spine, shoulder, knee, ankle, foot, hip (Musculoskeletal and connective tissue disorders) | 10 (10) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT03903874/Prot_SAP_000.pdf